CLINICAL TRIAL: NCT02095431
Title: Acute Kidney Injury Biomarkers: Diagnosis and Application in Pre-operative Period of Liver Transplantation
Acronym: AKIB
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Etienne Macedo, MD, PhD, University of Sao Paulo
Other Study IDs: 10393; 2013/12710-2 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2014-02-07; First posted 2014-03-24 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Acute Kidney Injury
Keywords: patients undergoing the liver transplantation; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasma and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- with AKI and without AKI: development of AKI by sCr and by novel biomarkers

SUMMARY:
Acute kidney injury (AKI), is a common complication of patients undergoing liver transplantation. Timing and definition of AKI, usually based on serum creatinine, have been inaccurate and inconsistent.

We hypothesized that the pattern of novel biomakers elevation could be a prognostic tool to provide information on the risk of progression of AKI, the need for RRT and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Reception liver transplantation

Exclusion Criteria:

* CKD stage 4 / 5
* Combined organ transplants
* Patients receiving dialysis before liver transplant operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to liver transplantation .
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Development of Acute Kidney Injury based on novel biomarkers | within 7 days
  Compare the timing for diagnosis of AKI comparing novel biomarkers and serum creatinine defined by Kidney Disease Improving Global Outcomes. In addition, we aim to evaluate if the pattern of elevation of the novel biomarkers provide information on progression and severity of AKI.

SECONDARY OUTCOMES:
Short and long term renal outcomes | 1 year
  renal function and need for RRT
Association of urine chemistry and microscopy to predict acute kidney injury | within 7 days of liver transplantation
  Association of urine chemistry and microscopy with novel biomarkers to predict AKI diagnosis and progression

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Macedo, MD, PhD, Principal Investigator — Faculty of Medicine, University of São Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Barri YM, Sanchez EQ, Jennings LW, Melton LB, Hays S, Levy MF, Klintmalm GB. Acute kidney injury following liver transplantation: definition and outcome. Liver Transpl. 2009 May;15(5):475-83. doi: 10.1002/lt.21682. PMID 19399734
- [Background] Feldkamp T, Bienholz A, Kribben A. Urinary neutrophil gelatinase-associated lipocalin (NGAL) for the detection of acute kidney injury after orthotopic liver transplantation. Nephrol Dial Transplant. 2011 May;26(5):1456-8. doi: 10.1093/ndt/gfr146. Epub 2011 Apr 12. No abstract available. PMID 21486868
- [Background] White LE, Hassoun HT. Inflammatory Mechanisms of Organ Crosstalk during Ischemic Acute Kidney Injury. Int J Nephrol. 2012;2012:505197. doi: 10.4061/2012/505197. Epub 2011 Jun 9. PMID 21826270
- [Background] Tsagalis G. Update of acute kidney injury: intensive care nephrology. Hippokratia. 2011 Jan;15(Suppl 1):53-68. PMID 21897760
- [Background] Macedo E, Mehta RL. Prerenal failure: from old concepts to new paradigms. Curr Opin Crit Care. 2009 Dec;15(6):467-73. doi: 10.1097/MCC.0b013e328332f6e3. PMID 19855270
- [Background] Nejat M, Pickering JW, Devarajan P, Bonventre JV, Edelstein CL, Walker RJ, Endre ZH. Some biomarkers of acute kidney injury are increased in pre-renal acute injury. Kidney Int. 2012 Jun;81(12):1254-62. doi: 10.1038/ki.2012.23. Epub 2012 Mar 14. PMID 22418979
- [Background] Sirota JC, Klawitter J, Edelstein CL. Biomarkers of acute kidney injury. J Toxicol. 2011;2011:328120. doi: 10.1155/2011/328120. Epub 2011 Oct 29. PMID 22131986
- [Background] Xu X, Ling Q, Wei Q, Wu J, Gao F, He ZL, Zhou L, Zheng SS. An effective model for predicting acute kidney injury after liver transplantation. Hepatobiliary Pancreat Dis Int. 2010 Jun;9(3):259-63. PMID 20525552
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Derived] Lima C, Santos Ferreira G, Vattimo MFF, de Paiva Haddad LB, Malbouisson LM, Carneiro D'Albuquerque LA, Maciel AT, Macedo E. Comprehensive biomarker assessment for predicting severe acute kidney injury and need of kidney replacement therapy in liver transplantation patients. Ren Fail. 2024 Dec;46(2):2402076. doi: 10.1080/0886022X.2024.2402076. Epub 2024 Sep 17. PMID 39287102
- [Derived] Lima C, de Paiva Haddad LB, de Melo PDV, Malbouisson LM, do Carmo LPF, D'Albuquerque LAC, Macedo E. Early detection of acute kidney injury in the perioperative period of liver transplant with neutrophil gelatinase-associated lipocalin. BMC Nephrol. 2019 Oct 15;20(1):367. doi: 10.1186/s12882-019-1566-9. PMID 31615452